CLINICAL TRIAL: NCT02806609
Title: Effect of Muscle Pain in Late Cold Water Immersion, Muscular Recruitment, Postural Control Dynamic and Sleep Quality in Soccer Athletes: Randomized Study and Blind
Brief Title: Effect of Muscle Pain in Late Cold Water Immersion, Muscular Recruitment, Postural Control Dynamic and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Christiane Macedo, First investigator, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COLD WATER IMMERSION
Record Dates: First submitted 2016-05-04; First posted 2016-06-20 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Pain; Sleep
Keywords: football; cryotherapy; balance; electromyography
MeSH Terms: conditions — Pain | interventions — WW Domain-Containing Oxidoreductase; Immersion; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Other): Cold water immersion, with 10 degrees, for 10 minutes
  Interventions: Other: Cold water immersion, with 10 degrees, for 10 minutes
- Group 2 (Other): immersion in water at room temperature
  Interventions: Other: immersion in water at room temperature
- Group 3 (Other): active recovery - running
  Interventions: Other: active recovery - running
- Group 4 (Other): rest in the chair
  Interventions: Other: rest in the chair

INTERVENTIONS:
Other: Cold water immersion, with 10 degrees, for 10 minutes — cold water immersion
  Arms: Group 1
Other: immersion in water at room temperature — immersion in water at room temperature
  Arms: Group 2
Other: active recovery - running — active recovery
  Arms: Group 3
Other: rest in the chair — rest in the chair
  Arms: Group 4

SUMMARY:
Objective: To evaluate the effect of cold water immersion in elayed onset muscle soreness, muscle recruitment, dynamic postural control and quality of sleep in young soccer players.

Methods: The sample will consist of 28 soccer players between 18 and 21 years of the same football club and with the same routine practices and games. At first athletes will respond to the IC and will be submitted to the test of a repetition maximum. After three days the athletes will analysis of muscle recruitment by electromyography and dynamic posture control through the force platform both during the time of shooting, moreover, will respond to scale the quality of sleep the previous night and one on pain, then they are instructed to perform a fatigue protocol for the quadriceps and then will be randomized to one of four intervention groups: cold water immersion, submersion in water at room temperature, or active recovery control. The same APPRAISAL be remade into three new moments, 24, 48 and 72 hours after the fatigue test.

Hypothesis: The variables will be considered: Pain intensity in the quadriceps muscle, quality of sleep the night after intervention protocol, electromyographic analysis of the rectus femoris, vastus medialis oblique and vastus lateralis at the time of shooting, as well as postural control when the shot off.

It is intended to establish the best way of recovery of late quadriceps muscle pain and contribute to the clinical practice of active recovery or rest in young soccer players.

DETAILED DESCRIPTION:
The size and power of the sample was raised with use of sample size calculation, the Power and Sample Size program with a 95% confidence interval, alpha level of 5% and power of 80%, considering the mean and standard deviation of data DOMS study the Effects of Cold Water Immersion after Rugby Training on muscle Power and Biochemical Markers. Thus, the sample was set at 48 volunteers, 12 distributed to each of the four groups.

Participate in the study 28 soccer players, aged between 16 and 21 years, male, with training at least 5 times a week, no complaints of musculoskeletal pain or history of muscle injuries in the past six months, hired a same club with the same demand for training and competitions.

Exclusion criteria will be observed vascular problems, allergy to cold, surgery of the lower limbs in the past six months, athletes in viral states (such as colds or flu).

These will be randomized into four groups: cold water immersion (N = 7) immersion in water at room temperature (n = 7), active recovery (n = 7) and control (N = 7).

ELIGIBILITY:
Inclusion Criteria:

* Soccer players
* Aged between 16 and 21 years
* Male
* Train at least 5 times a week
* No complaints of musculoskeletal pain or history of muscle injuries in the past six months
* Hired at the same club with the same demand for training and competitions

Exclusion Criteria:

* Exclusion criteria will be observed vascular problems
* Allergy to cold
* Surgery of the lower limbs in the past six months
* Athletes in viral states (such as colds or flu)

Ages: 16 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2016-06-01; Primary Completion 2016-12-30 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
visual pain scale | change of pain within 72 hours
  Demirhan et al. (2015) showed reduced muscle pain with the application of cold water immersion in elite wrestlers. Visual analogue range, ranging from 0 to 10, where 0 is no pain and 10 is maximum pain.

SECONDARY OUTCOMES:
balance by force platform | before the intervention and 24, 48 and 72 hours, by force platform
  Tano et al. (2015) did not establish differences in postural control after cryoimmune, but the results remain inconsistent.
muscle recruitment by electromyography | before the intervention and 24, 48 and 72 hours, by electromyography
  In a study carried out by Peter et al. (2015), CWI had no effects on the muscular response of physically active subjects. However, the assessment was performed immediately after the intervention, different from our study, which analyzed the effects of CWI immersion 72 hours after a DOMS-inducing protocol.
Sleep measured by Visual Analog Scale | before the intervention and 24, 48 and 72 hours, by questionnaire
  Robey et al. (2013) and Minet et al. (2015) found no effect of recovery methods on sleep quality of athletes. However, the relationship between sleep and performance has become a topic of great interest due to the growth of scientific evidence confirming the link between sleep and cognitive processes and metabolic functions in non-athletes. Spiegel's scale ranges from 1 to 5, where 5 means that he slept very well and 1 did not do well at all.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, doctor, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- Junior Football Team, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bleakley C, McDonough S, Gardner E, Baxter GD, Hopkins JT, Davison GW. Cold-water immersion (cryotherapy) for preventing and treating muscle soreness after exercise. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD008262. doi: 10.1002/14651858.CD008262.pub2. PMID 22336838
- [Background] Buchheit M, Peiffer JJ, Abbiss CR, Laursen PB. Effect of cold water immersion on postexercise parasympathetic reactivation. Am J Physiol Heart Circ Physiol. 2009 Feb;296(2):H421-7. doi: 10.1152/ajpheart.01017.2008. Epub 2008 Dec 12. PMID 19074671